CLINICAL TRIAL: NCT00253344
Title: Phase I Trial of Daily Lenalidomide (CC-5013, Revlimid™) and Docetaxel Given Every Three Weeks in Patients With Advanced Solid Tumors
Brief Title: Lenalidomide and Docetaxel in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Matthew Cooney, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2Y04; P30CA043703 (NIH); CASE2Y04 (Other: Case Comprehensive Cancer Center); AVENTIS-CASE-2Y04; CELGENE-CASE-2Y04
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Docetaxel; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel — Docetaxel IV over 1 hour on day 1. Courses repeat every 21 days until disease progression or unacceptable toxicity.
Drug: lenalidomide — Oral lenalidomide on days 1-14. Courses repeat every 21 days until disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with docetaxel may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lenalidomide when given together with docetaxel in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and maximum tolerated dose of lenalidomide when given in combination with docetaxel in patients with advanced solid tumors.

Secondary

* Determine the safety of this regimen in these patients.
* Determine the objective tumor response in patients treated with this regimen.
* Determine the time to progression in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of lenalidomide.

Patients receive oral lenalidomide on days 1-14 and docetaxel IV over 1 hour on day 1. Courses repeat every 21 days until disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of lenalidomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Advanced disease
  * Refractory to standard therapy OR no standard therapy exists
* Measurable or evaluable disease
* No active brain metastases

  * Previously treated (e.g., surgery or radiotherapy) brain metastases are allowed provided they are currently asymptomatic and inactive by CT scan or MRI

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* At least 4 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND AST or ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal

Renal

* Creatinine ≤ 2 mg/dL

Cardiovascular

* No New York Heart Association class III or IV heart disease

Immunologic

* No prior desquamating rash or ≥ grade 2 allergic reaction while receiving thalidomide
* No history of hypersensitivity to docetaxel or other drugs formulated in polysorbate 80
* No history of allergic reaction to compounds of similar chemical or biologic composition to study drugs

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other uncontrolled illness or other condition that would preclude study compliance
* No peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent hematopoietic growth factors during course 1 of study treatment
* No concurrent immunotherapy

Chemotherapy

* At least 6 weeks since prior mitomycin or nitrosoureas

  * No more than 2 prior courses of mitomycin
* No other concurrent chemotherapy

Radiotherapy

* No prior pelvic radiotherapy

Other

* At least 4 weeks since prior anticancer therapy
* No concurrent warfarin for anticoagulation (heparin is allowed)
* Recovered from all prior treatment
* No other concurrent anticancer therapy except bisphosphonates
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | measured at end of phase I
Dose-limiting toxicity | measured after every course

SECONDARY OUTCOMES:
Disease response | measured after every 2 courses

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M. Cooney, MD, Study Chair — Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Sanborn SL, Gibbons J, Krishnamurthi S, Brell JM, Dowlati A, Bokar JA, Nock C, Horvath N, Bako J, Remick SC, Cooney MM. Phase I trial of docetaxel given every 3 weeks and daily lenalidomide in patients with advanced solid tumors. Invest New Drugs. 2009 Oct;27(5):453-60. doi: 10.1007/s10637-008-9200-x. Epub 2008 Nov 15. PMID 19011760